CLINICAL TRIAL: NCT04260607
Title: Initiating Ketamine in Acutely Suicidal Patients in the Emergency Department
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As a busy MTF we were unable to retain a health care provider with the appropriate expertise to buy-in to this study once the initiating PI left military service.
Sponsor: Naval Medical Center Camp Lejeune (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMCCL.2018.0011
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Suicide; Suicide Threat; Depression Severe
Keywords: ketamine
MeSH Terms: conditions — Suicide | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Experimental versus Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple masked study (patient, healthcare provider, outcomes assessor) performed by pharmacy investigators not involved in study recruitment or assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental-Ketamine (Experimental): single dose IV Ketamine (Ketalar) 0.5mg/kg in 100ml Normal Saline infused over 40 minutes
  Interventions: Drug: Ketamine Hydrochloride
- Placebo-Saline (Placebo Comparator): 100ml Normal Saline infused over 40 minutes
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Experimental Procedure
  1. Baseline evaluation of suicidal severity (BSSI) & degree of depressive symptoms (MADRS-S) will be evaluated through self-administered questionnaires.
  2. The experimental and placebo arms will receive a single dose of IV ketamine, 0.5 mg/kg in 100 cc NS or 100 cc of NS infused over 40 minutes.
  3. Post ketamine re-evaluation of outcome measures at four and twenty-four hours will determine clinical effectiveness of ketamine intervention
  4. Inspection of admission and transfer time provides time measurement for LOS. This secondary measure is needed to determine efficiency of intervention.
  5. Post ketamine re-evaluation of outcome measure at one-week post infusion will elucidate ketamine's durability of effect.
  Other Names: Experimental Arm
  Arms: Experimental-Ketamine
Drug: Normal saline — Experimental Procedure
  1. Baseline evaluation of suicidal severity (BSSI) & degree of depressive symptoms (MADRS-S) will be evaluated through self-administered questionnaires.
  2. The placebo arms will receive a single dose of 100 cc of NS infused over 40 minutes.
  3. Post Placebo infusion re-evaluation of outcome measures at four and twenty-four hours
  4. Inspection of admission and transfer time provides time measurement for LOS. This secondary measure is needed to determine efficiency of intervention.
  5. Post Normal Saline re-evaluation of outcome measure at one-week post infusion.
  Other Names: Placebo Comparator
  Arms: Placebo-Saline

SUMMARY:
Current treatment for acutely suicidal patients are limited to hospitalization, psychotherapy, electro-convulsant therapy, or a combination of the aforementioned. However, this has added to the national boarding problem. Long term pharmacologic treatment for suicidal behaviors and mood stabilization has been studied in specific populations. In these populations, the decreases in suicidal ideation results from stabilization of the underlying psychiatric illness. Ketamine is most commonly used as an anesthetic with analgesic properties. It has been used off-label for pain management, procedural sedation, status epilepticus, and treatment resistant depression. It has been safely administered intravenously and well tolerated for chronic Post Traumatic Stress Disorder. It increases norepinephrine, dopamine, and serotonin through adrenergic neuron stimulation and prevention of catecholamine uptake. There is a strong corollary between stress and the development of depression and suicidal behaviors. It is proposed that the use of low dose intravenous ketamine may have benefit on the suicidal ideation of patients presenting to the Emergency Department.

DETAILED DESCRIPTION:
There is a strong corollary between stress and the development of depression and suicidal behaviors. The neurobiological mediators of stress are primarily controlled by the noradrenergic and corticotropin-releasing factor (CRF) median eminence systems. Furthermore, stress directly and indirectly, through the Hypothalamic Pituitary Axis, activates the Locus Coeruleus (LC), which is the primary producer of NE in the central nervous system (CNS). Directly, glutaminergic neurons send excitatory signals to the LC via interaction with N-Methyl-D-Aspartate (NMDA) receptors NMDA antagonists, such as ketamine, can dampen the glutaminergic system, which has been implicated during states of depression and low moods.

The neurobiological commonality between multiple psychiatric disorders and depression, suicide, and attempted suicide is a decrease in serotonergic activity. It has been shown that patients who died of suicide, have decreased serotonin transporter in the ventromedial prefrontal cortex and anterior cingulate, which are areas that control decision making or willful action. The prefrontal cortex is important for inhibitory behavioral control. A potential treatment modality of ketamine, is that it produces activation of this region.35 The anterior cingulate cortex has been shown to be associated with impulsive aggression compared to control. Clinical studies have shown that low CSF 5-HIAA, metabolite in serotonin system, has been implicated and positively correlated to aggression scores and impulsivity. This is interesting because, suicides in the military are thought to have an impulsivity component, triggered by one or more major life stressors.

Another region associated with suicide is the infralimbic cortex. A recent study, based on neuroimaging techniques, demonstrated that glucose metabolism in this region was associated with SI at baseline, and decreases in SI was observed after ketamine infusion. This is the same region target by deep brain stimulation, for depression treatment. Additionally, the infralimbic cortex has been implicated in behavioral flexibility. Implicating that ketamine's anti-suicidal properties may stem from its ability to promoting cognitive flexibility. Most likely due to its ability to increase brain-derived neurotrophic factor (BDNF), which is a major contributor to neuronal plasticity. BDNF also plays key roles in synaptic and long-term potentiation, which may counteract the decreased levels in Mood Disorder (MDD) patients. Furthermore, ketamine infusion has been shown to change sleep slow wave activity. This biomarker is functionally related to increased synaptic strengthening and cortical synchronization. These factors, combined, may be implicated in not only ketamine's antidepressant effects and counteraction of decreased synaptic plasticity seen mood disorders, but also its ability to have week long lasting effects.

This information leads us to hypothesize that treatment of acutely suicidal patients with ketamine would: 1) decrease suicidal ideationto a clinically significant degree, and 2) the effect of ketamine will be seen for as long as one-week post administration.

To the best of our knowledge, this study does not duplicate any ongoing work. Instead, it would strengthen power to past studies and current work. There are four clinical trials investigating ketamine's effect on SI. One has an unknown status. There are two that are investigating ketamine in relationship to psychiatric standard of care, whereas this study is investigating its effects against a saline placebo. Finally, the last clinical trial is investigating the Neurobiology of Suicide. Their phase 2 component, which utilizes a similar protocol, uses ketamine as a tool to identify potential biomarkers for suicide. Furthermore, this study differs from Janssen Research & Development's clinical trial in administration route and study design. Their study focuses on using ketamine through intranasal administration. Their primary outcomes are the long-term safety and efficacy, and the design of their study is an open label multicenter trial.

This research does not duplicate any prior work. To date, there is only one study, from Iran, that evaluates the effectiveness of ketamine in high risk patients, or those that present as acutely suicidal to the ED. This was a single blinded trial that utilized 0.2mg/kg infused over one minute. The study indicated significant decrease in their measurement outcomes. However, they concluded that ketamine is not a good choice for treatment because it did not meet their cut off values. Their results might have been influenced by the rapid infusion over one minute, which differs from our study as well as the vast majority of the literature. We believe the slower 40-minute infusion is necessary for optimal results, as the larger dosage has produced more clinically meaningful results in prior studies, and the slower infusion produced less negative side effects. They chose the minimal dose shown to diminish SI41 200 ng/ml (0.2 mg/kg), which provokes lateral nystagmus.35 This protocol utilizes a higher dose, 0.5 mg/kg, which is the ED50 for narcosis. Our study is medically relevant because dosage effects on SI have not been studied. Comparison of our studies may address questions regarding the optimal dose and infusion rate.

The BSSI will measure the severity of SI. It is based on the interviewer rated version of the original Scale for Suicidal Ideation (SSI), which is one of the few document suicide assessment tools with predictive validity for suicide completion. The internal reliability, test and retest validity, as well as invariance over time has been demonstrated for the BSS. Furthermore, the first five items of the BSSI are a common clinical screening for the presence of suicidal thoughts. For these reasons, the BSSI was chosen as our primary outcomes measure. Two studies have indicated that the cut off between high and low risk is a BSS ≥ 2. A recent investigation has determined BSSI ≥ 6 is predictive of future suicide attempts. These two values will serve in our analysis.

The Montgomery- Åsberg Depression Rating Scale (MADRS) is a widely known 10 item clinician administered measure of depression severity. Since it's development in the late 1970s, it has become more popular than the gold standard, Hamilton rating scale for Depression (HAM-D). It is considered to be more sensitive to change, just as effective, and simpler to use clinically. However, the reliability depends on good interrater agreement. Difficulties in clinical trial to show signal detection for known effective drugs have implicated clinician administered measurement as a possible source of error. To avoid poor interrater reliability, rater bias, and variable interview quality, this trial will utilize the self-administered version of the MADRS-S. This has 9 items and a total score ranging from 0 to 27.50 The scoring of MADRS-S has shown to be similar to that of physician scoring.

The emotional pain of the suicidal patient requires empathetic care that may not always be possible with the time pressures, volume, and pragmatic nature of the ED environment. A pharmacologic intervention with rapid effects to decrease SI would play a vital role in improving the standard of care for this vulnerable population.

ELIGIBILITY:
Subject Inclusion and Selection Criteria

1. Patient demographics will consist of Active, Reserve, or retired military personnel or their dependents.

   Subjects must meet the following inclusion criteria:
2. Adult (18 to 89 years old)
3. Present with active SI
4. Deemed to being admitted to inpatient psychiatric unit

Subject Exclusion Criteria:

1. Age < 18 years old or > 89 years old
2. Currently presenting with psychosis as determined by mental health consultant
3. Have a history of Cognitive disorder that would impair understanding of consent
4. Have a personal/family history of Schizophrenia
5. Currently pregnant or nursing
6. Serious and unstable medical condition/problems
7. Inability to medically clear
8. Non-English Speakers
9. Civilian Humanitarians
10. Have previously enrolled in this study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan H Butler, DO, Principal Investigator — Naval Medical Center Camp Lejeune
Locations (1):
- Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armed Forces Health Surveillance Center (AFHSC). Deaths by suicide while on active duty, active and reserve components, U.S. Armed Forces, 1998-2011. MSMR. 2012 Jun;19(6):7-10. PMID 22779434
- [Background] Owens PL, Fingar KR, Heslin KC, Mutter R, Booth CL. Emergency Department Visits Related to Suicidal Ideation, 2006-2013. 2017 Jan. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #220. Available from http://www.ncbi.nlm.nih.gov/books/NBK442036/ PMID 28722846
- [Background] Ting SA, Sullivan AF, Boudreaux ED, Miller I, Camargo CA Jr. Trends in US emergency department visits for attempted suicide and self-inflicted injury, 1993-2008. Gen Hosp Psychiatry. 2012 Sep-Oct;34(5):557-65. doi: 10.1016/j.genhosppsych.2012.03.020. Epub 2012 May 2. PMID 22554432
- [Background] Reinstatler L, Youssef NA. Ketamine as a potential treatment for suicidal ideation: a systematic review of the literature. Drugs R D. 2015 Mar;15(1):37-43. doi: 10.1007/s40268-015-0081-0. PMID 25773961
- [Background] Weiss AP, Chang G, Rauch SL, Smallwood JA, Schechter M, Kosowsky J, Hazen E, Haimovici F, Gitlin DF, Finn CT, Orav EJ. Patient- and practice-related determinants of emergency department length of stay for patients with psychiatric illness. Ann Emerg Med. 2012 Aug;60(2):162-71.e5. doi: 10.1016/j.annemergmed.2012.01.037. Epub 2012 May 2. PMID 22555337
- [Background] Hazlett SB, McCarthy ML, Londner MS, Onyike CU. Epidemiology of adult psychiatric visits to US emergency departments. Acad Emerg Med. 2004 Feb;11(2):193-5. PMID 14759965
- [Background] Baraff LJ, Janowicz N, Asarnow JR. Survey of California emergency departments about practices for management of suicidal patients and resources available for their care. Ann Emerg Med. 2006 Oct;48(4):452-8, 458.e1-2. doi: 10.1016/j.annemergmed.2006.06.026. Epub 2006 Aug 21. PMID 16997683
- [Background] Jick H, Kaye JA, Jick SS. Antidepressants and the risk of suicidal behaviors. JAMA. 2004 Jul 21;292(3):338-43. doi: 10.1001/jama.292.3.338. PMID 15265848
- [Background] Ribeiro JD, Gutierrez PM, Joiner TE, Kessler RC, Petukhova MV, Sampson NA, Stein MB, Ursano RJ, Nock MK. Health care contact and suicide risk documentation prior to suicide death: Results from the Army Study to Assess Risk and Resilience in Servicemembers (Army STARRS). J Consult Clin Psychol. 2017 Apr;85(4):403-408. doi: 10.1037/ccp0000178. PMID 28333538
- [Background] Betz ME, Wintersteen M, Boudreaux ED, Brown G, Capoccia L, Currier G, Goldstein J, King C, Manton A, Stanley B, Moutier C, Harkavy-Friedman J. Reducing Suicide Risk: Challenges and Opportunities in the Emergency Department. Ann Emerg Med. 2016 Dec;68(6):758-765. doi: 10.1016/j.annemergmed.2016.05.030. Epub 2016 Jul 21. PMID 27451339
- [Background] Betz ME, Boudreaux ED. Managing Suicidal Patients in the Emergency Department. Ann Emerg Med. 2016 Feb;67(2):276-82. doi: 10.1016/j.annemergmed.2015.09.001. Epub 2015 Oct 9. No abstract available. PMID 26443554
- [Background] Hickey L, Hawton K, Fagg J, Weitzel H. Deliberate self-harm patients who leave the accident and emergency department without a psychiatric assessment: a neglected population at risk of suicide. J Psychosom Res. 2001 Feb;50(2):87-93. doi: 10.1016/s0022-3999(00)00225-7. PMID 11274665
- [Background] Meltzer HY, Alphs L, Green AI, Altamura AC, Anand R, Bertoldi A, Bourgeois M, Chouinard G, Islam MZ, Kane J, Krishnan R, Lindenmayer JP, Potkin S; International Suicide Prevention Trial Study Group. Clozapine treatment for suicidality in schizophrenia: International Suicide Prevention Trial (InterSePT). Arch Gen Psychiatry. 2003 Jan;60(1):82-91. doi: 10.1001/archpsyc.60.1.82. PMID 12511175
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Wilkinson ST, Ballard ED, Bloch MH, Mathew SJ, Murrough JW, Feder A, Sos P, Wang G, Zarate CA Jr, Sanacora G. The Effect of a Single Dose of Intravenous Ketamine on Suicidal Ideation: A Systematic Review and Individual Participant Data Meta-Analysis. Am J Psychiatry. 2018 Feb 1;175(2):150-158. doi: 10.1176/appi.ajp.2017.17040472. Epub 2017 Oct 3. PMID 28969441
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Mion G, Villevieille T. Ketamine pharmacology: an update (pharmacodynamics and molecular aspects, recent findings). CNS Neurosci Ther. 2013 Jun;19(6):370-80. doi: 10.1111/cns.12099. Epub 2013 Apr 10. PMID 23575437
- [Background] Krupitsky EM, Burakov AM, Romanova TN, Grinenko NI, Grinenko AY, Fletcher J, Petrakis IL, Krystal JH. Attenuation of ketamine effects by nimodipine pretreatment in recovering ethanol dependent men: psychopharmacologic implications of the interaction of NMDA and L-type calcium channel antagonists. Neuropsychopharmacology. 2001 Dec;25(6):936-47. doi: 10.1016/S0893-133X(01)00346-3. PMID 11750186
- [Background] Mann JJ, Currier D. Medication in Suicide Prevention Insights from Neurobiology of Suicidal Behavior. In: Dwivedi Y, editor. The Neurobiological Basis of Suicide. Boca Raton (FL): CRC Press/Taylor & Francis; 2012. Chapter 21. Available from http://www.ncbi.nlm.nih.gov/books/NBK107195/ PMID 23035282
- [Background] Mann JJ, Currier DM. Stress, genetics and epigenetic effects on the neurobiology of suicidal behavior and depression. Eur Psychiatry. 2010 Jun;25(5):268-71. doi: 10.1016/j.eurpsy.2010.01.009. Epub 2010 May 6. PMID 20451357
- [Background] Mundt C, Reck C, Backenstrass M, Kronmuller K, Fiedler P. Reconfirming the role of life events for the timing of depressive episodes. A two-year prospective follow-up study. J Affect Disord. 2000 Jul;59(1):23-30. doi: 10.1016/s0165-0327(99)00127-5. PMID 10814767
- [Background] Skolnick P, Layer RT, Popik P, Nowak G, Paul IA, Trullas R. Adaptation of N-methyl-D-aspartate (NMDA) receptors following antidepressant treatment: implications for the pharmacotherapy of depression. Pharmacopsychiatry. 1996 Jan;29(1):23-6. doi: 10.1055/s-2007-979537. PMID 8852530
- [Background] Scheuch K, Holtje M, Budde H, Lautenschlager M, Heinz A, Ahnert-Hilger G, Priller J. Lithium modulates tryptophan hydroxylase 2 gene expression and serotonin release in primary cultures of serotonergic raphe neurons. Brain Res. 2010 Jan 11;1307:14-21. doi: 10.1016/j.brainres.2009.10.027. Epub 2009 Oct 17. PMID 19840776
- [Background] Bowdle TA, Radant AD, Cowley DS, Kharasch ED, Strassman RJ, Roy-Byrne PP. Psychedelic effects of ketamine in healthy volunteers: relationship to steady-state plasma concentrations. Anesthesiology. 1998 Jan;88(1):82-8. doi: 10.1097/00000542-199801000-00015. PMID 9447860
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Schloesser RJ, Huang J, Klein PS, Manji HK. Cellular plasticity cascades in the pathophysiology and treatment of bipolar disorder. Neuropsychopharmacology. 2008 Jan;33(1):110-33. doi: 10.1038/sj.npp.1301575. Epub 2007 Oct 3. PMID 17912251
- [Background] Price RB, Mathew SJ. Does ketamine have anti-suicidal properties? Current status and future directions. CNS Drugs. 2015 Mar;29(3):181-8. doi: 10.1007/s40263-015-0232-4. PMID 25715884
- [Background] Kashani P, Yousefian S, Amini A, Heidari K, Younesian S, Hatamabadi HR. The Effect of Intravenous Ketamine in Suicidal Ideation of Emergency Department Patients. Emerg (Tehran). 2014 Winter;2(1):36-9. PMID 26495340
- [Background] Brown GK, Beck AT, Steer RA, Grisham JR. Risk factors for suicide in psychiatric outpatients: a 20-year prospective study. J Consult Clin Psychol. 2000 Jun;68(3):371-7. PMID 10883553
- [Background] van Spijker BA, Majo MC, Smit F, van Straten A, Kerkhof AJ. Reducing suicidal ideation: cost-effectiveness analysis of a randomized controlled trial of unguided web-based self-help. J Med Internet Res. 2012 Oct 26;14(5):e141. doi: 10.2196/jmir.1966. PMID 23103835
- [Background] de Beurs DP, Fokkema M, de Groot MH, de Keijser J, Kerkhof AJ. Longitudinal measurement invariance of the Beck Scale for Suicide Ideation. Psychiatry Res. 2015 Feb 28;225(3):368-73. doi: 10.1016/j.psychres.2014.11.075. Epub 2014 Dec 23. PMID 25571773
- [Background] Asberg M, Montgomery SA, Perris C, Schalling D, Sedvall G. A comprehensive psychopathological rating scale. Acta Psychiatr Scand Suppl. 1978;(271):5-27. doi: 10.1111/j.1600-0447.1978.tb02357.x. No abstract available. PMID 277059
- [Background] Khan A, Khan SR, Shankles EB, Polissar NL. Relative sensitivity of the Montgomery-Asberg Depression Rating Scale, the Hamilton Depression rating scale and the Clinical Global Impressions rating scale in antidepressant clinical trials. Int Clin Psychopharmacol. 2002 Nov;17(6):281-5. doi: 10.1097/00004850-200211000-00003. PMID 12409681
- [Background] Muller MJ, Szegedi A. Effects of interrater reliability of psychopathologic assessment on power and sample size calculations in clinical trials. J Clin Psychopharmacol. 2002 Jun;22(3):318-25. doi: 10.1097/00004714-200206000-00013. PMID 12006903
- [Background] Bondolfi G, Jermann F, Rouget BW, Gex-Fabry M, McQuillan A, Dupont-Willemin A, Aubry JM, Nguyen C. Self- and clinician-rated Montgomery-Asberg Depression Rating Scale: evaluation in clinical practice. J Affect Disord. 2010 Mar;121(3):268-72. doi: 10.1016/j.jad.2009.06.037. Epub 2009 Aug 5. PMID 19660815
- [Background] Bartoli F, Riboldi I, Crocamo C, Di Brita C, Clerici M, Carra G. Ketamine as a rapid-acting agent for suicidal ideation: A meta-analysis. Neurosci Biobehav Rev. 2017 Jun;77:232-236. doi: 10.1016/j.neubiorev.2017.03.010. Epub 2017 Mar 23. PMID 28342764
- [Background] de Beurs DP, Fokkema M, O'Connor RC. Optimizing the assessment of suicidal behavior: The application of curtailment techniques. J Affect Disord. 2016 May 15;196:218-24. doi: 10.1016/j.jad.2016.02.033. Epub 2016 Feb 23. PMID 26938964
- [Background] Zarate CA Jr, Brutsche N, Laje G, Luckenbaugh DA, Venkata SL, Ramamoorthy A, Moaddel R, Wainer IW. Relationship of ketamine's plasma metabolites with response, diagnosis, and side effects in major depression. Biol Psychiatry. 2012 Aug 15;72(4):331-8. doi: 10.1016/j.biopsych.2012.03.004. Epub 2012 Apr 18. PMID 22516044
- [Background] Khan A, Brown WA. The placebo enigma in antidepressant clinical trials. J Clin Psychopharmacol. 2001 Apr;21(2):123-5. doi: 10.1097/00004714-200104000-00001. No abstract available. PMID 11270906
- [Background] Monteggia LM, Zarate C Jr. Antidepressant actions of ketamine: from molecular mechanisms to clinical practice. Curr Opin Neurobiol. 2015 Feb;30:139-43. doi: 10.1016/j.conb.2014.12.004. Epub 2015 Jan 3. PMID 25562451
- [Background] Nagels A, Kirner-Veselinovic A, Wiese R, Paulus FM, Kircher T, Krach S. Effects of ketamine-induced psychopathological symptoms on continuous overt rhyme fluency. Eur Arch Psychiatry Clin Neurosci. 2012 Aug;262(5):403-14. doi: 10.1007/s00406-011-0281-8. Epub 2011 Dec 22. PMID 22189657
- [Background] Hartvig P, Valtysson J, Lindner KJ, Kristensen J, Karlsten R, Gustafsson LL, Persson J, Svensson JO, Oye I, Antoni G, et al. Central nervous system effects of subdissociative doses of (S)-ketamine are related to plasma and brain concentrations measured with positron emission tomography in healthy volunteers. Clin Pharmacol Ther. 1995 Aug;58(2):165-73. doi: 10.1016/0009-9236(95)90194-9. PMID 7648766
- [Background] Strayer RJ, Nelson LS. Adverse events associated with ketamine for procedural sedation in adults. Am J Emerg Med. 2008 Nov;26(9):985-1028. doi: 10.1016/j.ajem.2007.12.005. PMID 19091264
- [Background] Clattenburg EJ, Hailozian C, Haro D, Yoo T, Flores S, Louie D, Herring AA. Slow Infusion of Low-dose Ketamine Reduces Bothersome Side Effects Compared to Intravenous Push: A Double-blind, Double-dummy, Randomized Controlled Trial. Acad Emerg Med. 2018 Sep;25(9):1048-1052. doi: 10.1111/acem.13428. Epub 2018 May 25. PMID 29645317
- See also: Violence Prevention [Internet]. Centers for Disease Control and Prevention, National Center for Injury Prevention and Control, 2018 [cited 2018 July 1]. — https://www.cdc.gov/injury
- See also: Medical care of the returning veteran. Up To Date. — https://www.uptodate.com/contents/medical-care-of-the-returning-veteran?topicRef=1708&source=see_link.
- See also: Knesper DJ. Continuity of care for suicide prevention and research: Suicide attempts and suicide deaths subsequent to discharge from the emergency department or psychiatry inpatient unit. 2010. Newton, MA: Suicide Prevention Resource Center. 68(6):758- — https://sprc.org/wp-content/uploads/2022/11/continuityofcare.pdf
- See also: Ketamine. Lexicomp; 31 January 2020. — https://online.lexi.com/lco/action/doc/retrieve/docid/patch_f/7135?cesid=3kjMrqmcjDs&searchUrl=%2Flco%2Faction%2Fsearch%3Fq%3Dketamine%26t%3Dname%26va%3Dketamine
- See also: Janssen Research & Development, LLC. A Long-term, Safety and Efficacy study of Intranasal Esketamine in Treatment resistant depression (SUSTAIN-2). 2017. ClinicalTrials.gov. — https://clinicaltrials.gov/ct2/show/record/NCT02497287?view=record
- See also: Neurobiology of Suicide. 2018. ClinicalTrials.Gov. — https://clinicaltrials.gov/ct2/show/record/NCT02543983?view=record.
- See also: Pearson, 2018. Administering the Beck Scale Suicidal Ideation® (BSS®) Via Telepractice. — https://www.pearsonclinical.com/RelatedInfo/telepractice/telepractice-and-the-bss.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruitment occurred from main ED from 2019-2021
Pre-assignment Details: Medical Record review completed
Groups:
- Experimental-Ketamine: single dose IV Ketamine (Ketalar) 0.5mg/kg in 100ml Normal Saline infused over 40 minutes
  Ketamine Hydrochloride: Experimental Procedure
  1. Baseline evaluation of suicidal severity (BSSI) & degree of depressive symptoms (MADRS-S) will be evaluated through self-administered questionnaires.
  2. The experimental and placebo arms will receive a single dose of IV ketamine, 0.5 mg/kg in 100 cc NS or 100 cc of NS infused over 40 minutes.
  3. Post ketamine re-evaluation of outcome measures at four and twenty-four hours will determine clinical effectiveness of ketamine intervention
  4. Inspection of admission and transfer time provides time measurement for LOS. This secondary measure is needed to determine efficiency of intervention.
  5. Post ketamine re-evaluation of outcome measure at one-week post infusion will elucidate ketamine's durability of effect.
- Placebo-Saline: 100ml Normal Saline infused over 40 minutes
  Normal saline: Experimental Procedure
  1. Baseline evaluation of suicidal severity (BSSI) & degree of depressive symptoms (MADRS-S) will be evaluated through self-administered questionnaires.
  2. The placebo arms will receive a single dose of 100 cc of NS infused over 40 minutes.
  3. Post Placebo infusion re-evaluation of outcome measures at four and twenty-four hours
  4. Inspection of admission and transfer time provides time measurement for LOS. This secondary measure is needed to determine efficiency of intervention.
  5. Post Normal Saline re-evaluation of outcome measure at one-week post infusion.
Period: Overall Study
Arm/Group | Experimental-Ketamine | Placebo-Saline
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As a busy MTF we were unable to retain a health care provider with the appropriate expertise to buy-in to this study once the initiating PI left military service. At the time the PI left military service, only 1 patient had been assigned to the experimental group, and 0 patients to the placebo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental-Ketamine | Placebo-Saline | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: Years] | 23 [23 to 23] |  | 23 [23 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Beck Scale for Suicide Ideation (BSS) [Median (Full Range); unit: units on a scale] — The BSS is a self-administered 21-item scale. Each item contains a group of statements that are rated from 0 to 2. Items 1 to 5 comprise a screening subscale. If the patient scores 0 in total on items 4 and 5, items 6 to 19 are skipped. Item 21 is only asked if the patient has attempted suicide at least once. A high total score corresponds with an increased number of specific suicidal characteristics that require greater clinical scrutiny.
  units on a scale
    Screening Subscore | 7 [7 to 7] |  | 7 [7 to 7]
    Total Score | 29 [29 to 29] |  | 29 [29 to 29]
Montgomery Asberg Depression Rating Scale (MADRS) [Median (Full Range); unit: units on a scale] — Depression symptoms are measured by the total score on the Montgomery Asberg Depression Rating Scale (MADRS). The MADRS is a self-administered questionnaire that consists of 9 items. Each item is scored between 0 and 3, in intervals of 0.5 The total scores range between 0 and 27, with higher scores indicating more severe depressive symptoms.
  units on a scale | 20 [20 to 20] |  | 20 [20 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Suicidal Severity - Clinical Efficacy
Description: Suicidal severity is measured by the total score on the Beck Scale for Suicide Ideation (BSS or BSSI). The BSS is a 21-item scale, where each item contains a group of statements that are rated from 0 to 2. Items 1 to 5 comprise a screening subscale. If the patient scores 0 in total on items 4 and 5, items 6 to 19 are skipped. Item 21 is only asked if the patient has attempted suicide at least once. The screening subscale can range from 0 to 10 points, whereas the total score can range from 0 to 42 points. A high total score corresponds with an increased number of specific suicidal characteristics that require greater clinical scrutiny.
Time Frame: 4 hour+/1 after infusion completion (performed for placebo and drug arms)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 1 | 0
Units on a Scale | 3 [3 to 3] |

2. Primary Outcome: Suicidal Severity - Clinical Efficacy
Description: as for outcome 1
Time Frame: 24-36 hours after infusion completion (performed for placebo and drug arms)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 1 | 0
Units on a Scale | 2 [2 to 2] |

3. Primary Outcome: Suicidal Severity - Efficacy at 1 Week
Description: as for outcome 1
Time Frame: 1week+/-1 day after infusion completion (performed for placebo and drug arms)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 1 | 0
Units on a Scale | 6 [6 to 6] |

4. Primary Outcome: Depression Symptoms - Clinical Efficacy
Description: Depression symptoms are measured by the total score on the Montgomery Asberg Depression Rating Scale (MADRS). The MADRS scale consists of 9 items. Each item is scored between 0 and 3, in intervals of 0.5 The total scores range between 0 and 27, with higher scores indicating more severe depressive symptoms.
Time Frame: 4 hours +/-1 after infusion completion (Performed for placebo and drug arms)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 1 | 0
units on a scale | 7 [7 to 7] |

5. Primary Outcome: Depression Symptoms - Clinical Efficacy
Description: as for outcome 4
Time Frame: 24-46 hours after infusion completion (Performed for placebo and drug arms)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 1 | 0
units on a scale | 2 [2 to 2] |

6. Primary Outcome: Depression Symptoms - Efficacy at 1 Week
Description: as for outcome 4
Time Frame: 1 week +/-1 day after infusion completion, performed for placebo and drug arms
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 1 | 0
units on a scale | 9.5 [9.5 to 9.5] |

7. Secondary Outcome: Length of Hospital Stay
Description: Difference in time between date of hospital admission to transfer or hospital discharge.
Time Frame: Performed on medical record review at 1 week
Population: The length of hospital stay was not recorded for the patient.
Arm/Group | Experimental-Ketamine | Placebo-Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: N/A; Definition of adverse event and/or serious adverse event, is the same as the clinicaltrials.gov definition.
Arm/Group | Experimental-Ketamine | Placebo-Saline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental-Ketamine (N=1) | Placebo-Saline (N=0)
Mild Severity AE (Psychiatric disorders) | 1 (1) | NA — Subject hearing voices when subject goes to sleep at night Study intervention relationship possibly related, but expected.

LIMITATIONS AND CAVEATS:
As a busy MTF we were unable to retain a health care provider with the appropriate expertise to buy-in to this study once the initiating PI left military service. At the time the PI left military service, only one patient had been assigned to the experimental group, and 0 patients to the placebo group. While data from the one patient was reported in the results with descriptive statistics, no inferential analysis could be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT04260607/Prot_SAP_002.pdf
  • Informed Consent Form (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04260607/ICF_001.pdf